CLINICAL TRIAL: NCT00306982
Title: An Observational Study to Investigate the Incidence of Influenza, Downstream Complications of Influenza and Hospitalizations, in Elderly Subjects Vaccinated With GSK Biologicals' Influenza Vaccine (Fluarix™) Administered Intramuscularly.
Brief Title: Incidence of Influenza, Downstream Complications of Influenza & Hospitalizations in Elderly Vaccinated With Fluarix™
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 106622
Record Dates: First submitted 2006-02-27; First posted 2006-03-27 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Influenza
Keywords: Prophylaxis Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Biological: Fluarix

SUMMARY:
This study will investigate the incidence of influenza, disease and various possible downstream complications and hospitalizations or emergency room visits after routine annual vaccination of the elderly population with Fluarix™.

DETAILED DESCRIPTION:
This study will investigate the incidence of influenza, disease and various possible downstream complications, such as pneumonia, ischemic HD (unstable angina or MI), congestive heart failure, acute cerebrovascular disease, COPD exacerbation and hospitalizations or emergency room visits, and will evaluate the feasibility of health outcome surveillance and the validity of using questionnaires instruments, after routine annual vaccination of the elderly population with Fluarix™.

ELIGIBILITY:
Inclusion Criteria

All subjects must satisfy to the following criteria at study entry:

* (1) A male or female age 65 years at the time of the first vaccination,
* (2) Subjects who the investigator believes that they can and will comply with the requirements of the protocol (e.g., return for follow-up visits, disease reporting by phone, and completion of Questionnaires) should be enrolled in the study
* (3) Written informed consent obtained from the subject
* (4) Availability to follow up by phone during the study period
* (5) Subjects with residence status allowing free mixing with general community.

Exclusion Criteria

The subject must not be included in the study for:

* (1) history of hypersensitivity to a previous dose of influenza vaccine
* (2) history of allergy or reactions likely to be exacerbated by any component of the vaccine including egg, chicken protein, formaldehyde, thimerosal, gentamicin sulfate or sodium deoxycholate,
* (3) use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 1524 (Actual)
Dates: Start 2006-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Australia (10):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Umina, New South Wales
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, South Brisbane, Queensland
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Clayton, Victoria
  - GSK Investigational Site, Heidelberg Heights, Victoria
  - GSK Investigational Site, Parkville, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Brazil (2):
  - GSK Investigational Site, Curitiba/Paraná, Paraná
  - GSK Investigational Site, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106622 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register